CLINICAL TRIAL: NCT02574143
Title: The PROspective German NOn-CF bronchiectaSIS Patient Registry
Acronym: PROGNOSIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: CAPNETZ Stiftung (Other); German Center for Lung Research (Other)
Responsible Party: Sponsor
Other Study IDs: PROGNOSIS
Record Dates: First submitted 2015-07-17; First posted 2015-10-12 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Bronchiectasis
Keywords: Prognosis; Prospective Study; Quality of Life; Radiology; Rehabilitation; Registry;; Signs and Symptoms; Therapy; Bronchiectiasis; Diagnosis; Epidemiology; Etiology; Longitudinal Study; Microbiology
MeSH Terms: conditions — Bronchiectasis; Signs and Symptoms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the epidemiology of non-CF bronchiectasis (NCFB) and to provide an estimate of the distribution (prevalence) of NCFB etiologies across all different levels of health care as well as real-life data regarding the current management of NCFB in Germany.

DETAILED DESCRIPTION:
* To study the epidemiology of non-CF bronchiectasis (NCFB) and to provide an estimate of the distribution (prevalence) of NCFB etiologies across all different levels of health care as well as real-life data regarding the current management of NCFB in Germany
* To establish feasible investigational strategies in order to establish the etiology of NCFB
* To perform observational research into bronchiectasis, particularly in areas where single center datasets are underpowered, such as in rare etiologies or determining markers of prognosis
* To promote collaborative clinical, basic and translational research in NCFB between German (and European) centers
* To provide a registry of well phenotyped patients with NCFB in clinical centers potentially eligible for enrolment into clinical trials
* To track access to healthcare and cost of caring for patients with NCFB over time

ELIGIBILITY:
Inclusion Criteria:

* A clinical history consistent with bronchiectasis
* (High resolution) computed tomography (CT) scan of the chest demonstrating bronchiectasis affecting 1 or more lobes

Exclusion Criteria:

* Bronchiectasis due to known cystic fibrosis (CF)
* Age <18 years
* Interstitial lung disease
* Prior lung or heart-lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-CF bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-11 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-CF bronchiectasis (NCFB) across all different levels of health care regarding the current management of NCFB in Germany | three years
  To establish a national, representative, prospective, observational and longitudinal NCFB database and collaborative research network with a database including a minimum of 750 patients from a minimum of 25 centers from all levels of healthcare across Germany after a period of 3 years.

SECONDARY OUTCOMES:
Prevalence of non-CF bronchiectasis (NCFB) etiologies (composite outcome measures) across all different levels of health care | three years
  * Distribution (prevalence) of underlying conditions/etiologies
  * Clinical presentation of NCFB
  * Predictors of lung function decline in patients with NCFB
  * Diagnostics employed in determining the etiology of NCFB
  * Microbiology of NCFB
  * Radiology of NCFB
  * Comorbidity in patients with NCFB
  * Impact of exacerbations and hospitalizations on the clinical course of NCFB
  * Prescription patterns of pharmacological respiratory treatments for NCFB
  * Usage and benefit of surgical procedures in NCFB
  * Physical therapy and rehabilitation
  * Healthcare utilization and associated costs in NCFB
  * QOL(Questions of Life) among patients with NCFB
  * survival/mortality of NCFB

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rademacher, Study Chair — CAPNETZ STIFTUNG; Medizinische Hochschule Hannover; Felix C. Ringshausen, Study Chair — CAPNETZ STIFTUNG; Medizinische Hochschule Hannover; Andrés de Roux, Study Chair — Pneumologische Praxis Berlin
Locations (19):
- Germany (19):
  - Helios Klinikum Emil von Behring - Lungenklinik Heckeshorn, Berlin
  - Augusta-Kranken-Anstalt Bochum -Klinik für Pneumologie, Beatmungsmedizin und Infektiologie, Bochum
  - Fachkrankenhaus Coswig, Coswig
  - Klinik Donaustauf - Zentrum für Pneumologie, Donaustauf
  - Klinikum Dortmund Medizinische Klinik Nord - Pneumologie, Infektiologie und Internistische Intensivmedizin, Dortmund
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden Medizinische Klinik und Poliklinik I, Bereich Pulmologie, Dresden
  - Florence-Nightingale-Krankenhaus Klinik für Pneumologie, Allergologie, Schlaf- und Beatmungsmedizin, Düsseldorf
  - Praxis am Maingau Krankenhaus Gemeinschaftspraxis für Innere Medizin, Lungen- und Bronchialheilkunde, Allergologie, Frankfurt
  - Universitätsklinikum Freiburg Abteilung für Klinische Infektiologie, Freiburg im Breisgau
  - UKGM - Standort Gießen Medizinische Klinik und Poliklinik II, Giessen
  - LungenClinic Großhansdorf, Großhansdorf
  - Medizinische Hochschule Hannover-Klinik für Pneumologie, Hanover
  - Universitätsklinikum Heidelberg und Thoraxklinik Heidelberg, Heidelberg
  - Universitätsklinikum Jena Zentrum für Infektionsmedizin und Krankenhaushygiene, Jena
  - Universitätsklinikum Schleswig-Holstein Medizinische Klinik III - Pneumologie / Infektiologie, Lübeck
  - Klinikum Lüdenscheid Klinik für Pneumologie, Infektiologie, Schlafmedizin und Internistische Intensivmedizin, Lüdenscheid
  - Klinikum der Philipps-University Marburg, Marburg
  - Klinikum der Ludwig-Maximilians-Universität München, München
  - Diakoniekrankenhaus Rotenburg Zentrum für Pneumologie, Rotenburg (Wümme)

REFERENCES:
- [Derived] Ewen R, Pink I, Sutharsan S, Aries SP, Grunewaldt A, Shoemark A, Sommerwerck U, Staar BO, Wege S, Mertsch P, Rademacher J, Ringshausen FC; PROGNOSIS Study Group. Primary Ciliary Dyskinesia in Adult Bronchiectasis: Data from the German Bronchiectasis Registry PROGNOSIS. Chest. 2024 Nov;166(5):938-950. doi: 10.1016/j.chest.2024.05.023. Epub 2024 Jun 15. PMID 38880279
- See also: PROGNOSIS - das deutsche Bronchiektasen-Register — http://www.bronchiektasen-register.de